CLINICAL TRIAL: NCT01297569
Title: An Open-label, Prospective, Multicentre, Uncontrolled, Proof of Concept Study Assessing the Efficacy of Lucentis (Ranibizumab) Administered by an Individualized "Treat and Extend" Dosing Regimen in Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: Ranibizumab "Treat and Extend" in Diabetic Macular Edma
Acronym: OPTIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DNO02; 2010-021182-76 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Macular edema; DME; Diabetic retinopathy; Diabetic eye disease; anti-VEGF; ranibizumab; Lucentis
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — Ranibizumab

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
This study is designed to explore a more individualized treatment regime based on achievement of disease stability to define a personal optimal treatment interval with ranibizumab in patients with visual impairment due to diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment due to focal or diffuse macular edema with center involvement
* Diabetes type 1 or 2, HbA1c < 12.0%
* CRT = or > 250 μm

Exclusion Criteria:

* Active inflammation or infection
* Uncontrolled glaucoma
* Iris neovascularization, active proliferative retinopathy or vitreomacular traction
* Prior laser photocoagulation according to defined timelines
* History of stroke, uncontrolled hypertension

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity(BCVA) | from month 0 (baseline) to month 12

SECONDARY OUTCOMES:
change in central retinal thickness (CRT) | from month 0 to month 12
the number of injections needed | 12 months
the number of patients with improvement in BCVA from baseline | 12 months
the number of patients with > 5, 10 and 15 letters improvement from baseline, the latter including patients reaching BCVA >84 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Oslo, Norway